CLINICAL TRIAL: NCT03237767
Title: A CFit Study: To What Extent Does a Single Session of Exercise Training Influence Measures of Inflammation, Oxidative Stress, Nitric Oxide Bioavailability, Microvascular Endothelial Function and Dysglycaemia in Patients With Cystic Fibrosis?
Brief Title: A CFit Study - Acute Exercise
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: University of Portsmouth (Other)
Collaborators: Queen Alexandra Hospital, Portsmouth (Unknown); University Hospital Southampton NHS Foundation Trust (Other); Loughborough University (Other)
Responsible Party: Principal Investigator, Dr Zoe Saynor, Senior Lecturer in Physical Activity, Exercise and Health, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZS003
Record Dates: First submitted 2017-07-26; First posted 2017-08-03 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis-related Diabetes
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: The present study will be a pilot, counter-balanced, cross-over trial in individuals with CF.
Masking Description: The present study will be a pilot, counter-balanced, cross-over trial in individuals with CF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate vs. High-intensity exercise (randomised) (Experimental): Compare the effects of a single session of moderate continuous exercise versus high-intensity interval exercise (MIE completed first)
  Interventions: Other: MIE; Other: HIIE
- High-intensity vs. Moderate intensity exercise (randomised) (Experimental): Compare the effects of a single session of moderate continuous exercise versus high-intensity interval exercise (HIIE completed first)
  Interventions: Other: MIE; Other: HIIE

INTERVENTIONS:
Other: MIE — The moderate intensity exercise (MIE) condition will begin and end with an appropriate warm-up (3 minutes at 20 W) and cool-down (2 minutes at 20 W), respectively. Throughout all exercising procedures, participants will maintain a pedal cadence of 60-80 rpm, with the average being noted and kept consistent between trials. Additionally, verbal encouragement will be given depending on the participant's preference, and kept consistent between visits.
  The MIE bout will be in coherence with the physical activity guidelines for people with CF (150 min/week of moderate to vigorous physical activity). For the MIE, participants will cycle for approximately 30 minutes at 90% of their gas exchange threshold.
Other: HIIE — The high-intensity interval exercise (HIIE) condition will begin and end with an appropriate warm-up (3 minutes at 20 W) and cool-down (2 minutes at 20 W), respectively. Throughout all exercising procedures, participants will maintain a pedal cadence of 60-80 rpm, with the average being noted and kept consistent between trials. Additionally, verbal encouragement will be given depending on the participant's preference, and kept consistent between visits.
  The HIIE will be matched for the projected work done during the MIE. The HIIE protocol has been extrapolated from recent reports which have shown improvements in glycaemic control and vascular endothelial function. Specifically, participants will cycle at 90% of their peak power output for 60 seconds, followed by 60 seconds of active recovery.

SUMMARY:
A great medical success is the increase in the median survival age associated with cystic fibrosis (CF). However, this success has led to a new era of research aiming to maximise the quality of life (QoL) of the aging CF population. Over recent decades, exercise training has become an integral part of CF management by improving ones aerobic exercise function and QoL. However, the effects exercise training has upon other aspects of the disease, e.g. metabolic and vascular abnormalities, remains largely unknown.

The increased survival age associated with CF means the non-pulmonary co-morbidities are becoming increasingly prevalent and clinically important. For example, CF-related diabetes (CFRD) is one of the most common non-pulmonary co-morbidities of CF, and is associated with patients having a poorer pulmonary function and nutritional state, which ultimately leads to a worsened prognosis. Despite the efficacy of exercise training to manage dysglycaemia in other populations (e.g. type 2 diabetes mellitus only a single study has investigated its efficacy in patients with CF, whereby authors reported various encouraging findings (e.g. an improved OGTT score and insulin sensitivity).

The present study aims to build on previous trials by comparing the therapeutic effects of a single session of high-intensity interval exercise (HIIE) and moderate intensity exercise (MIE) upon the 24 hour, ambulatory glycaemic profile of patients with CF. Additionally, the present study will identify whether HIIE and/or MIE can mediate the consequences of transient hyperglycaemia when considering: biomarkers of inflammation, oxidative stress and nitric oxide (NO2) bioavailability, as well as functional measures of microvascular endothelial function.

The present study supports the top 10 research priorities set by the CF Trust, by further investigating the potential for exercise training to prevent/manage multiple aspects of CF, including dysglycaemia.

DETAILED DESCRIPTION:
Participants and recruitment The present study will be a pilot, counter-balanced, cross-over trial in individuals with CF (n = 16). Furthermore, the present protocol is an extension of the CFit_BL protocol (Clinical Trials ID to be confirmed). Specifically, 16 participants with CF will be invited to complete 2 visits (5 in total) within the same 14 day time period. Briefly, participants will be recruited from adult and paediatric CF outpatient clinics within the Southampton CF network, and will be tested at a laboratory within the Southampton General Hospital or the Department of Sport and Exercise Sciences (University of Portsmouth), depending on participant convenience.

The present study will comprise 2 visits which will be in a randomised, counter-balanced order.

Visits 1 and 2 A session of moderate intensity exercise (MIE) training and high-intensity interval exercise (HIIE) training visit will be conducted in a randomised, counter-balanced order. Participants will be required to arrive to the laboratory ~ 96 hours following the previous visit, at 0800 ± 2 hours, following an overnight fast (> 10 hours). Furthermore, participants will be instructed to avoid nitrate rich foods, caffeine, alcohol and exhaustive exercise for 24 hours prior to arrival, as well as mouthwash for the entirety of the study.

Upon arrival, CGM's will be fixed to the interior surface of the upper arm and worn for the subsequent 14 days. In addition to this, hip worn accelerometers, as well as hourly specific physical activity and food diaries will be distributed and completed for 14 days alongside the CGM.

Upon arrival participants will undergo the acetylcholine (ACh) and insulin iontophoresis protocols described below, including 5 resting blood pressure measurements and a cannula will be inserted into a vein by a trained phlebotomist, prior to the 3 hour OGTT and a baseline blood sample will be taken. The participant's pulmonary function will be assessed via spirometry. Participants will then be asked to complete either a single session of either MIE or HIIE.

Pulmonary function will then be assessed immediately post-exercise. 1 hour following exercise, the iontophoresis procedures will be repeated. Blood samples will be drawn immediately pre- and post-exercise for the analysis of plasma TNF-α, soluble vascular cell adhesion molecule (sVCAM)-1, IL-6, [NO-(₂)] and ET-1. Samples for nitrotyrosine (NT), total glutathione (tGSH) and total cysteine (tCys) will be drawn pre-exercise only. Subsequently, participants will partake in either 30 minutes of MIE or a work-matched period of HIIE. Thirty minutes following the completion of the exercising procedures, the iontophoresis procedures will be repeated and blood samples will be drawn for the analysis of plasma glucose, insulin, TNF-α, sVCAM-1, IL-6, [NO-(₂)] and ET-1. NT, tGSH and tCys. Following this, 1.75 g/kg body mass (maximum of 75 g) of anhydrous glucose will be consumed to instigate the 3 hour OGTT, whereby blood samples will be drawn at 30, 60, 90, 120 and 180 minutes post-glucose ingestion for the analysis of glucose and insulin. Samples for TNF-α, sVCAM-1, IL-6, [NO-(₂)] and ET-1 will be drawn at 60, 120 and 180 minutes post-glucose ingestion. NT, tGSH and tCys will be analysed at 120 minutes post-glucose ingestion. The total volume of blood collected over each 5 hour visit will be approximately 232 mL. Additionally, the iontophoresis procedures will be repeated at 30, 90 and 150 minutes post-glucose ingestion.

Follow-up CGM's, accelerometers and physical activity/food diaries will be completed throughout this 14 day period. A member of the research team will collect these from the preferred location of the participant.

ELIGIBILITY:
Inclusion Criteria:

* Males and females ≥ 12 years of age
* CF diagnosis based on clinical features, supported by an abnormal sweat test (sweat chloride > 60 mmol·L-1 > 100 mg sweat) and, where possible, diagnostic genotyping
* No contraindications to performing exhaustive exercise
* Can understand and cooperate with the study protocol
* No increase in symptoms or weight loss in the preceding 2 weeks

Exclusion Criteria:

* Any non-pulmonary conditions that may impair exercise ability, such as musculoskeletal disorders (arthritis, joint or muscle disease) and cardiovascular disease (congenital heart disease or cardiomyopathy).
* Unstable co-morbid asthma (daily pulmonary function variability of > 20%)
* Is pregnant during the initial screening process
* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Not of a suitable age for testing

Exclusion during testing:

* Onset of acute infection
* Becomes and/or is tested to be pregnant following enrolment to the study
* Experiences significant hypoxaemia during visit 2 of the CFit_BL protocol (IRAS ID: 225310) which requires supplemental O₂. Under these circumstances, participants will be invited to continue their participation under the CFit_BL trial (IRAS ID: 225310)
* Unable to understand or cooperate with study protocol
* The individual does not wish to participate further

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Glucose concentration before and after oral glucose tolerance test | Visit 1 (pre glucose ingestion after exercise completed and 30, 60, 90, 120 and 180 minutes following glucose ingestion), Visit 2 (pre glucose ingestion after exercise completed and 30, 60, 90, 120 and 180 minutes following glucose ingestion)
  Glucose concentration before and after oral glucose tolerance test (which follows an exercise training session)
Insulin concentration before and after oral glucose tolerance tolerance | Visit 1 (pre glucose ingestion after exercise completed and 30, 60, 90, 120 and 180 minutes following glucose ingestion), Visit 2 (pre glucose ingestion after exercise completed and 30, 60, 90, 120 and 180 minutes following glucose ingestion)
  Insulin concentration before and after oral glucose tolerance test (which follows an exercise training session)
Glycaemic control (measured using arm-mounted Freestyle Libre continuous glucose monitor) | Continuous measurement through study completion (2 week period)
  Glycaemic control fixed to the arm will measure glucose excursions continuously

SECONDARY OUTCOMES:
Nitrotyrosine (NT) | Visit 1 and 2: pre-exercise (baseline) and 1 h following exercise 75 g glucose is ingested: NT measured immediately before glucose ingestion and 120 minutes after
  Nitrotyrosine (NT) measured from plasma
Total cysteine (tCys) | Visit 1 and 2: pre-exercise (baseline) and 1 h following exercise 75 g glucose is ingested: tCys measured immediately before glucose ingestion and 120 minutes after
  Total cysteine (tCys) measured from plasma
Total glutathione (tGSH) | Visit 1 and 2: pre-exercise (baseline) and 1 h following exercise 75 g glucose is ingested: tGSH measured immediately before glucose ingestion and 120 minutes after
  Total glutathione (tGSH) measured from plasma
Tumor necrosis factor alpha (TNF-alpha) | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: TNF-alpha measured immediately before glucose ingestion and 60, 120 and 180 minutes after)
  Tumor necrosis factor alpha (TNF-alpha) measured from plasma
Soluble vascular cell adhesion molecule (sVCAM-1) | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: sVCAM-1 measured immediately before glucose ingestion and 60, 120 and 180 minutes after)
  Soluble vascular cell adhesion molecule-1 (sVCAM-1) measured from plasma
Endothelin-1 (ET-1) | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: ET-1 measured immediately before glucose ingestion and 60, 120 and 180 minutes after)
  Endothelin-1 (ET-1)
Interleukin-6 (IL-6) | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: IL-6 measured immediately before glucose ingestion and 60, 120 and 180 minutes after)
  Interleukin-6 (IL-6)
[Nitrite] ([NO2]) | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: NO2 measured immediately before glucose ingestion and 60, 120 and 180 minutes after)
  [Nitrite] ([NO2])measured from plasma
Pulmonary function (forced expiratory volume in 1 second, forced vital capacity, peaf expiratory flow and mid-forced expiratory flow) measured using flow-volume loop spirometry | Visit 1 and 2: pre-exercise (baseline) and immediately post-exercise, additionally 1 h following exercise 75 g glucose is ingested: pulmonary function measured immediately before glucose ingestion
  Pulmonary function will be measured using flow-volume spirometry and presented in both absolute units and as a percentage of predictive normative reference values
Insulin iontophoresis | Visit 1 and 2: pre-exercise (baseline), additionally 1 h following exercise 75 g glucose is ingested: insulin iontophoresis measured immediately before glucose ingestion and 1, 2 and 3 hours after.
  Insulin iontophoresis measures of microvascular endothelial function
Acetylcholine iontophoresis | Visit 1 and 2: pre-exercise (baseline), additionally 1 h following exercise 75 g glucose is ingested: acetylcholine iontophoresis measured immediately before glucose ingestion and 1, 2 and 3 hours after.
  Acetylcholine iontophoresis measures of microvascular endothelial function
Dietary intake | Continuous measurement through study completion (2 weeks), participants will record everything that they eat and drink
  Dietary intake measured using MyFitness Pal application and dietary records
Physical activity | Continuous measurement through study completion (2 week period)
  Physical activity measured using wrist worn accelerometer (GeneActiv)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will be shared with the research team only.